CLINICAL TRIAL: NCT04297839
Title: Evaluation of the Efficacy and Safety of Regional Anticoagulation With Citrate in Extended Hemodialysis in Patients With Acute Renal Injury Admitted to an Intensive Care Unit
Brief Title: Evaluation of Regional Anticoagulation With Citrate in Extended Hemodialysis
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: DUE TO CORONAVIRUS DISEASE, ACTIVITIES INTHE HOSPITAL ARE SUPRESSED
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other); Hospital do Cancer, Sao Paulo (Other)
Responsible Party: Principal Investigator, EMMANUEL DE ALMEIDA BURDMANN, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6293
Record Dates: First submitted 2019-10-28; First posted 2020-03-06 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Hemodialysis Complication; Acute Kidney Injury; Anticoagulant Toxicity
Keywords: Extended Hemodialysis; Anticoagulation; Citrate; Heparin; Coagulation in Dialysis
MeSH Terms: conditions — Acute Kidney Injury | interventions — Citric Acid; Control Groups; Heparin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Open label randomized clinical trial with cross-over between the groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (Active Comparator): Patients in this group will receive heparin during hemodialysis sessions, at a dose of 1.000 units at the beginning and 500 units per hour in a syringe infusion pump.
  If the patient has a contraindication for the heparin use, it will receive saline continuous administration.
  This is the actual standard of care performed in extended hemodialysis sessions.
  Interventions: Drug: Control Group (heparin or continuous saline)
- Citrate Group (Experimental): Patients in this group will receive regional citrate anticoagulation, with acid-citrate-dextrose 2.2% (ACD). Dose of 3 mmol per liter of filtered blood. The systemic calcium levels are measured every two hours and a solution of calcium chloride is infused in a peripheral venous access, accordingly to citrate infusion rate and the systemic calcium values.
  Interventions: Drug: Citrate Anticoagulation Solution

INTERVENTIONS:
Drug: Citrate Anticoagulation Solution — Regional citrate anticoagulation in extended hemodialysis sessions compared to the standard of care actually performed in these therapies (heparin or continuous saline infusion)
  Other Names: Citrate
  Arms: Citrate Group
Drug: Control Group (heparin or continuous saline) — Use of heparin in hemodialysis sessions. If there is any contraindication against the use of heparina, the investigators will perform saline flush of the dialysis system
  Other Names: Heparin; Saline
  Arms: Control Group

SUMMARY:
Data on regional citrate anticoagulation in patients with acute kidney injury (AKI) treated by hybrid or extended dialysis are scarce and heterogeneous. The path batch system (Genius®) or the proportion hemodialysis machines are well suited equipments to perform extended dialysis. However, clotting of the system might occur with relatively high frequency, especially in critically ill patients with high risk of clotting or in those with contraindication to the use of heparin.

The aims of this study are: 1) to test and to validate a new protocol using citrate to perform regional anticoagulation in AKI patients admitted to the intensive care unit (ICU) and treated by extended dialysis, using a control group (use of heparin or intermittent saline flush) as comparison in the Heart Institute of the university medical complex "Clinics Hospital Medical School at São Paulo" (Hospital das Clínicas da Faculdade de Medicina do Estado de São Paulo) and at the Cancer Institute of the São Paulo State; 2) to evaluate the anticoagulation in these procedures with citrate and compare with the control group using heparin or saline flush, so the primary end point would be the rates of system clotting; 3) to study the calcium mass transfer in these procedures and its impact on bone metabolism in these patients. The inclusion criteria are all AKI patients admitted in these places and candidates to renal replacement therapy using the extended dialysis, age above 18 years. The exclusion criteria are acute liver failure, hemorrhagic stroke, platelets level below 20,000/mm3, and active bleeding needing transfusional support (two or more red cell packs in 24 hours).

DETAILED DESCRIPTION:
The investigators conduct an open label randomized clinical trial with cross-over between the groups. The study will be performed in all the intensive care units (ICU) at the Heart Institute and the Cancer Institute, both hospitals related with the University of São Paulo Medical School, at the city of São Paulo, Brazil.

All inpatients over 18 years in the ICU with acute kidney injury (AKI) who are arranged for extended hemodialysis will be invited to participate in the study. After signing an informed consent formulary, the patients went to randomization between two groups: citrate or control therapy. The research team randomly drawn the patients using a box with twenty entries for each group, totalizing forty units. Thus, after the inclusion of forty patients, it is guaranteed that half of them will start in the citrate group and the other half in the control group. Afterwards, the box is refilled to its maximum capacity of forty units for the next draw.

The randomization process determine the type of anticoagulation that the patient will be submitted in the first dialysis session. Subsequently the subject will participate in the other group, alternating between the two modalities until the maximum of six extended dialysis for the protocol.

In the control group, the decision on the use of heparin or continuous saline infusion as an anticoagulation method will be based on the presence of contraindications to the heparin use, which would be I) platelet levels <150,000/mm3; II) active or recent bleeding; III) reduction in hemoglobin levels of more than 2.0g/dl in less than 24 hours; IV) invasive procedures or surgeries realized in the last 7 days or scheduled to the next 24 hours.

There may be a change in the choice of method (citrate versus control), if the nephrologist consultant team deems it necessary, due to demands of care, particularly if there is early or repeated coagulation of the system. The proper functioning of the hemodialysis catheter will be evaluated before the dialysis initiation, and in case of malfunction, it will be properly replaced before the procedure starts.

The study foresees the inclusion of 800 dialytic procedures. Half of them are expected to be performed in the citrate group and half in the control group. As each patient can perform up to six procedures, it is estimated that approximately 200 patients will participate in this study. Data in the other intermittent dialysis not included in this trial and performed in the intensive care setting during the same period will be registered.

Patients will be excluded if they present: I) acute liver failure; II) hemorrhagic stroke in the last 30 days; III) platelet levels below 20,000/mm3 and IV) active bleeding requiring transfusion of two or more red blood cell packs within 24 hours.

Decisions about the need for renal replacement therapy, modality and time will be made by the nephrologist attendant. Intermittent methods are preferred performed in stable patients with no vasoactive drug, or with low doses of these drugs (norepinephrine <0.2 mcg/kg/min and dobutamine <5 mcg/kg/min).

All slow extended dialysis (SLED) in this trial were performed in 6 to 8 hours using a single-pass batch machine (Genius 90 Therapy System® Fresenius Medical Care, Bad Homburg, Germany), initiated by a nephrology specialized nurse and managed by an exclusive attendant. In this device, blood and dialysate flow rates are equal and set in 180 ml/min. We used only high-flux polysulfone filter (Ultraflux® AV 600S, Fresenius Medical Care). In the SPB device, the dialysate is stored in an air-free 90 liters glass container (batch system). Dialysate solution after proper reconstitution has sodium 138 mEq/l, bicarbonate 32.6 mEq/l, magnesium 1.0 mEq/l, chloride 111 mEq/l, potassium 2.0 or 3.0 mEq/l and calcium 2.5 mEq/l (5.0 mg/dl). Dialysate temperature was set in 36-37°C.

Citrate dose was tailored to achieve 3 mmol per filtered blood liter using a citric acid solution 2.2% 800 ml bag (each 100 mL of the solution contains 730 mg of citric acid, 2.45 g of dextrose and 2.2g of sodium citrate). Calcium replacement began if the patient has a serum ionized calcium less than 4.4 mg/dl (or 1.10 mmol/l) before it starts or during the session. We obtained blood samples at every two hours to adjust the calcium infusion rate targeting serum calcium from 4.4 to 5.3 mg/dl (or 1.10 to 1.32 mmol/l), using a calcium solution with 10% calcium chloride solution (concentration at 0.133 mmol/ml). The post filter ionized calcium addressed was 2.4 to 2.8 mg/d (or 0.6 to 0.7 mmol/l). Furthermore, in the control group, the equipment receive continuous saline in a infusion rate of 180 ml per hour or unfractionated heparin 1,000 units in bolus at the initiation of the procedure and maintained at 500 units per hour in a specific syringe pump in the device.

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute kidney injury admitted to the intensive care unit and candidates for extended dialysis (renal replacement therapy)
* Age over 18 years.

Exclusion Criteria:

* Acute liver failure
* Hemorrhagic stroke in the last 30 days
* Patients with platelet levels below 20,000/mm3
* Active bleeding requiring transfusion (two or more red blood cell packs within 24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Clotting rate | through all dialysis session, an average of 8 hours
  Clotting of the dialysis system with complete impossibility to continue the therapy

SECONDARY OUTCOMES:
Parathyroid hormone (PTH), Fibroblast growth factor-23 (FGF-23), Procollagen type 1 N-terminal propeptide (P1NP), Esclerostin and Telopeptide carboxiterminal of type I collagen (cTX) | through all dialysis session, an average of 8 hours
  Serum hormone levels will be evaluated before the dialysis session
Dialysate calcium | through all dialysis session, an average of 8 hours
  Dialysate calcium will be evaluated to address the calcium balance
Serum ionized and total calcium levels | through all dialysis session, an average of 8 hours
  Measurement before and after the dialysis session. In the citrate group it will be measured every 2 hours.
Serum sodium concentration | through all dialysis session, an average of 8 hours
  Measurement before and after the dialysis session. In the citrate group it will be measured every 2 hours.
Serum potassium concentration | through all dialysis session, an average of 8 hours
  Measurement before and after the dialysis session. In the citrate group it will be measured every 2 hours.
Serum bicarbonate | through all dialysis session, an average of 8 hours
  Measurement before and after the dialysis session. In the citrate group it will be measured every 2 hours.
Serum phosphorus | through all dialysis session, an average of 8 hours
  Measurement before and after the dialysis session.
Serum magnesium | through all dialysis session, an average of 8 hours
  Measurement before and after the dialysis session.
Serum creatinine concentration | through all dialysis session, an average of 8 hours
  Measurement before and after the dialysis session.
Serum urea concentration | through all dialysis session, an average of 8 hours
  Measurement before and after the dialysis session.
Parathyroid hormone (PTH) concentration | two measurements per patient (before the dialysis initiation and at the end, after an average of 8 hours)
  Serum hormone levels will be evaluated before the dialysis session
Fibroblast growth factor-23 (FGF-23) concentration | baseline, before the dialysis initiation
  Serum hormone levels will be evaluated before the dialysis session
Procollagen type 1 N-terminal propeptide (P1NP) concentration | baseline, before the dialysis initiation
  Serum hormone levels will be evaluated before the dialysis session
Sclerostin concentration | baseline, before the dialysis initiation
  Serum hormone levels will be evaluated before the dialysis session
Telopeptide carboxyterminal of type I collagen (cTX) concentration | baseline, before the dialysis initiation
  Serum hormone levels will be evaluated before the dialysis session
Mean arterial pressure | every hour in the dialysis session (an average of 8 hours)
  Patients in dialysis will have their blood pressure recorded every hour
Heart rate | every hour in the dialysis session (an average of 8 hours)
  Patients in dialysis will have their heart rate recorded every hour
Respiratory rate | every hour in the dialysis session (an average of 8 hours)
  Patients in dialysis will have their respiratory rate recorded every hour
Temperature | every hour in the dialysis session (an average of 8 hours)
  Patients in dialysis will have their temperature rate recorded every hour

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo Medical School, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The researchers have hot decided yet about this issue